CLINICAL TRIAL: NCT02743572
Title: Efficacy and Safety of Parenteral Nutrition With Iron Sucrose for Anemia in Preterm Infants: a Randomized, Double-blind Controlled Study
Brief Title: Iron-fortified Parenteral Nutrition in the Prevention and Treatment of Anemia in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, qingya tang, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: XH-16-002
Record Dates: First submitted 2016-03-31; First posted 2016-04-19 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Premature Birth
Keywords: premature infant; anemia; iron-fortification; parenteral nutrition; randomized controlled trial
MeSH Terms: conditions — Premature Birth; Anemia; Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- control group (No Intervention): preterm infants of this group with iron-free PN for more than seven days, compare erythrocyte parameters, serum iron, iron protein and MDA on baseline and after intervention
- iron sucrose-1 (Experimental): preterm infants of this group with iron supplementation of 100μg/kg/d for more than seven days, compare erythrocyte parameters, serum iron, iron protein and MDA on baseline and after intervention
  Interventions: Other: iron sucrose-1
- iron sucrose-2 (Experimental): preterm infants of this group with iron supplementation of 200μg/kg/d for more than seven days, compare erythrocyte parameters, serum iron, iron protein and MDA on baseline and after intervention
  Interventions: Other: iron sucrose-2
- iron sucrose-3 (Experimental): preterm infants of this group with iron supplementation of 300μg/kg/d for more than seven days, compare erythrocyte parameters, serum iron, iron protein and MDA on baseline and after intervention
  Interventions: Other: iron sucrose-3
- iron sucrose-4 (Experimental): preterm infants of this group with iron supplementation of 400μg/kg/d for more than seven days, compare erythrocyte parameters, serum iron, iron protein and MDA on baseline and after intervention
  Interventions: Other: iron sucrose-4

INTERVENTIONS:
Other: iron sucrose-1 — iron sucrose-1 group with PN of iron supplementation of 100μg/kg/d
  Arms: iron sucrose-1
Other: iron sucrose-2 — iron sucrose-2 group with PN of iron supplementation of 200μg/kg/d
  Arms: iron sucrose-2
Other: iron sucrose-3 — iron sucrose-3 group with PN of iron supplementation of 300μg/kg/d
  Arms: iron sucrose-3
Other: iron sucrose-4 — iron sucrose-4 group with PN of iron supplementation of 400μg/kg/d
  Arms: iron sucrose-4

SUMMARY:
The purpose of this study is to determine whether iron-fortified PN is effective in the preventative and treatment of preterm infants. Preterm infants are at risk for anemia especially in preterm infants. Anemia effects growing development, clinical prognosis, cognition, movement, learning ability and behavioral development.

As enteral nutrition is not feasible soon after birth in most preterm infants, parenteral iron administration is an efficacious method for investigators to select. For most preterm infants, the use of parenteral nutrition(PN) is very common during the first ten days of life, so the investigators hypothesis that iron-fortified PN may have a preventative and treatment effect on preterm infants using PN as a supplementation of oral nutrition; Iron-fortified PN can also improve iron store status of preterm infants. The higher concentration of iron used in this study, the larger preventative or treatment effect on preterm infants anemia; it is safe to add small dose of iron agent to PN.

DETAILED DESCRIPTION:
Infants are at risk for anemia especially in preterm infants. Generally the smaller birth weight and gestational age, the higher anemia ate in infants. As enteral nutrition is not feasible soon after birth in most preterm infants, parenteral iron administration is an efficacious method for investigators to select.

Meeting the Inclusion Criteria of this study will be randomly divided into five groups, control group, group1 (100μg/kg/d, and the highest concentration of iron is ≤0.8g/100ml PN), group2（200μg/kg/d, and the highest concentration of iron is ≤0.8g/100ml PN), group3 (300μg/kg/d, and the highest concentration of iron is ≤0.8g/100ml PN), group4 (400μg/kg/d, and the highest concentration of iron is ≤0.8g/100ml PN). Iron supplementation period for more than ten days. For five groups, complete blood counts, differential counts, and reticulocyte counts were measured weekly in samples obtained, serum iron, iron protein, total iron binding force were measured at baseline and after 2 weeks. Through comparative analysis of five groups, to find iron-fortified PN whether affect anemia rate and iron storage in premature infants. The investigators also selected malondialdehyde (MDA) and 8-isoprostaglandin F2α (8-iso-PGF2α) as the investigators concerns about iron used in PN induces oxidative stress index. Iron protein determination use radioimmunoassay method, serum iron and total iron binding force determination use chemical method, MDA and 8-iso-PGF2α determination use enzyme-linked immunosorbent assay method.

The investigators hypothesis that iron-fortified PN may have a preventative and treatment effect on preterm infants using PN as a supplementation of parenteral nutrition; Iron-fortified PN can also improve iron store status of preterm infants. The higher concentration of iron used in this study, the larger preventative or treatment effect on preterm infants anemia.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with birth weight less than 2kg
* Have parenteral nutrition indication
* With written informed consent of parents or guardian

Exclusion Criteria:

* Have already used PN before randomization
* Kidney and liver function abnormal
* Have hemolytic disease
* Have hemorrhagic disease
* Have Serious congenital malformation
* Have septicemia
* Have plethora newborn
* Use PN less than ten days

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes of iron status index before and after iron-fortified parenteral nutrition support | up to 2 weeks

SECONDARY OUTCOMES:
Changes of iron storage index before and after iron-fortified parenteral nutrition support | up to 1 month

OTHER OUTCOMES:
Changes of oxidative stress index before and after iron-fortified parenteral nutrition support | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: qingya tang, Principal Investigator — Shanghai jiaotong university affiliated xinhua hospital
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang S, Zeng L, Brouwer ID, Kok FJ, Yan H. Effect of iron deficiency anemia in pregnancy on child mental development in rural China. Pediatrics. 2013 Mar;131(3):e755-63. doi: 10.1542/peds.2011-3513. Epub 2013 Feb 11. PMID 23400604
- [Result] Singh S, Singh S, Singh PK. A study to compare the efficacy and safety of intravenous iron sucrose and intramuscular iron sorbitol therapy for anemia during pregnancy. J Obstet Gynaecol India. 2013 Mar;63(1):18-21. doi: 10.1007/s13224-012-0248-3. Epub 2012 Sep 12. PMID 24431594
- [Result] Inder TE, Clemett RS, Austin NC, Graham P, Darlow BA. High iron status in very low birth weight infants is associated with an increased risk of retinopathy of prematurity. J Pediatr. 1997 Oct;131(4):541-4. doi: 10.1016/s0022-3476(97)70058-1. PMID 9386655
- [Result] Cooke RW, Drury JA, Yoxall CW, James C. Blood transfusion and chronic lung disease in preterm infants. Eur J Pediatr. 1997 Jan;156(1):47-50. doi: 10.1007/s004310050551. PMID 9007491
- [Result] Moshtaghie M, Malekpouri P, Dinko MR, Moshtaghie AA. Changes in serum parameters associated with iron metabolism in male rat exposed to lead. J Physiol Biochem. 2013 Jun;69(2):297-304. doi: 10.1007/s13105-012-0212-9. Epub 2012 Sep 25. PMID 23007736
- [Result] Smith S. Safe administration of intravenous iron therapy. Nurs Stand. 2013 Apr 3-9;27(31):45-8. doi: 10.7748/ns2013.04.27.31.45.e5162. PMID 23641637
- [Result] Plummer ES, Crary SE, McCavit TL, Buchanan GR. Intravenous low molecular weight iron dextran in children with iron deficiency anemia unresponsive to oral iron. Pediatr Blood Cancer. 2013 Nov;60(11):1747-52. doi: 10.1002/pbc.24676. Epub 2013 Jul 6. PMID 23832487
- [Result] Heming N, Letteron P, Driss F, Millot S, El Benna J, Tourret J, Denamur E, Montravers P, Beaumont C, Lasocki S. Efficacy and toxicity of intravenous iron in a mouse model of critical care anemia*. Crit Care Med. 2012 Jul;40(7):2141-8. doi: 10.1097/CCM.0b013e31824e6713. PMID 22564959